CLINICAL TRIAL: NCT05439070
Title: Is Urdu Version of Northwick Park Neck Pain Questionnaire a Culturally Adaptable and Valid Tool to Assess the Neck Pain in Pakistani Population?
Brief Title: Urdu Version of Northwick Park Neck Pain Questionnaire: Reliability and Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00269
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Neck Pain
Keywords: Northwick Park Neck Pain Questionnaire; Urdu Version; Reliability; Validity; Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* To adapt culturally Neck Pain Questionnaire in Urdu language.
* To check the reliability of Urdu version of Neck Pain Questionnaire
* To validate Neck Pain Questionnaire by Neck Disability Index and Visual Analogue Scale and Numeric Pain Rating Scale.

DETAILED DESCRIPTION:
The original English version of Northwick Park Neck Pain Questionnaire will be translated and culturally adapted as per previous recommendation. In patients with neck pain, Urdu Version of Northwick Park Neck Pain Questionnaire will be distributed among 70 participants choose a convenience sampling technique based on pre-defined inclusion and exclusion criteria. To test reliability of inter/intra observer of ultimate final Urdu Version of Northwick Park Neck Pain Questionnaire will be filled from patients on the equivalent day, by 2 different bystanders, and for inter observer valuation, with an interval of 30 minutes between the first and second application. Third assessment will be carried out after 7 days of the Observer -1, for intra-observer assessment. Data will be entered and analyzed Cronbach alpha value. Test-retest reliability will be assessed using an intraclass correlation coefficient. Urdu Version of Northwick Park Neck Pain Questionnaire will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Both Male and Female
2. Minimum age is 18 years
3. Maximum age up to 60 years
4. People with Chronic neck pain
5. Duration of pain more then 3 months
6. No history of neck therapy
7. Not had any neck therapy

Exclusion Criteria:

1. People with medical history regarding skeleton issues
2. People with traumas
3. Having Neck surgery
4. People with neurological deficits ( like malignancies or inflammatory arthritis)
5. People went for therapy were also excluded.
6. People with age more than 60 and less than 18 were excluded..

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People suffering from chronic neck pain with a working routine of more than 3 to 4 both in sitting and standing position.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Northwick Park Neck Pain Questionnaire | 1st day
  Each parameter of Northwick Park Neck Pain Questionnaire has divided into 5 answers with total of 10 parameters. Each parameter is divided in five answer possibilities with points from 0 till 4. 0 is significant for no pain and 4 is significant for worst pain.
Neck Disability Index | 1st day
  Neck Disability Index includes ten questions that assess pain intensity, personal care, lifting, reading, headaches, attention, work, driving, sleeping, and recreational activities. Every question is graded on a scale of 0 to 5 (no disability to total disability).
Visual Analogue Scale | 1st day
  The Visual Analogue Scale was created to represent the concept of a fundamental continuity. A Visual Analogue Scale is typically a straight stripe measuring 100 mm long, with word descriptions for each end. The patient draws a line through the spot on the line which they believe best describes their present state. The Visual Analogue Scale score is calculated by calculating in millimeters as from the line's left side to the point marked by that of the patient. It usually ranges from "0" indicating "no pain" to the "10" indicating "worst pain".
Numeric Pain Rating Scale | 1st day
  Numeric Pain Rating Scale has a line value ranging from 1 to 10, 1 being the no pain label and 10 being the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No